CLINICAL TRIAL: NCT05376423
Title: A Randomized, Open-Label, Phase 2 Study to Evaluate Adjuvant OBI-833/OBI-821 Therapy in Patients With Locally Advanced, Globo H-Positive Esophageal Cancer at High Risk for Recurrence
Brief Title: To Evaluate OBI-833/OBI-821 in Patients With Locally Advanced, Globo H-Positive Esophageal Cancer for Recurrence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202106018MIPB
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OBI-833/OBI-821 (Experimental): OBI-833 consists of Globo H, a unique tumor-associated carbohydrate antigen (TACA), covalently linked to cross-reacting material 197 (CRM197), an inactive and nontoxic form of diphtheria toxin (DT) acting as a carrier protein.
  OBI-821 is a purified saponin adjuvant
  Dosage form: solution Dosage:30 μg OBI-833/100 μg OBI-821, subcutaneous injection, Frequency: weekly for 4 doses (weeks 1, 2, 3, 4), then every 2 weeks for 2 doses (weeks 6, 8), then every 4 weeks for 4 doses (weeks 12, 16, 20, 24), and then every 8 weeks until disease recurrence, intolerable adverse events/toxicity, consent withdrawal, death, or up to 80 weeks from randomization.
  Interventions: Biological: OBI-833/OBI-821
- Observation (No Intervention): Patients will be randomized into OBI-833/OBI-821 (experimental) arm or observation arm.

INTERVENTIONS:
Biological: OBI-833/OBI-821 — OBI-833 and OBI-821 are individually formulated into separate glass vials. The articles are mixed prior to subcutaneous administration at the clinic.
  Arms: OBI-833/OBI-821

SUMMARY:
A Phase 2 Study to Evaluate Adjuvant OBI-833/OBI-821 Therapy in Patients With Locally Advanced, Globo H-Positive Esophageal Cancer at High Risk for Recurrence

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, 20 years of age or older at the time of consent.
2. Pathologically or cytologically confirmed diagnosis of esophageal cancer (including squamous cell carcinoma and adenocarcinoma) whose postneoadjuvant pathologic stage is ypT1-4 AND ypN1-3 according to the AJCC Cancer Staging System, 8th Edition.
3. Patients have been treated with preoperative cisplatin-based chemoradiotherapy followed by esophagectomy with lymph node dissection for locally advanced esophageal cancer (defined by the above criterion).
4. Postneoadjuvant pathologic staging: ypT1-4 and ypN1-3.
5. Globo H IHC H-score ≥1 in the surgical tumor specimen from the primary site/or lymph node (if the primary site is not available). The Globo H expression will be determined by a qualified laboratory.
6. R0 (no residual tumor on the surgical margin of the resected tumor specimen).
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. Organ Function Requirements - Subjects must have adequate organ functions as defined below:

   * AST/ALT ≤ 3X ULN (upper limit of normal)
   * Total bilirubin ≤ 2X ULN
   * Serum creatinine ≤ 1.5X ULN
   * ANC ≧ 1,500 /μL
   * Platelets ≧ 100,000/μL
9. All eligible patients of childbearing potential must use effective contraception during study treatment and for at least 2 months after the last dose of OBI-833/OBI-821. Subjects not of childbearing potential (i.e., permanently sterilized, postmenopausal) can be included in the study. Postmenopausal is defined as 12 months with no menses without an alternative medical cause.
10. Ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria:

1. Subjects who cannot be randomized within 8 weeks after the esophageal cancer surgery.
2. Subjects who are pregnant or breast-feeding at entry.
3. Subjects with splenectomy.
4. Has prior malignancy, except (a) adequately treated basal cell or squamous cell skin cancer; (b) in situ cervical cancer; (c) previously diagnosed malignancy which has been adequately treated and shown no evidence of recurrence for more than 5 years.
5. Subjects with HIV infection, active hepatitis B infection, or active hepatitis C infection.
6. Subjects with any autoimmune or other disorders requiring IV/oral steroids or immunosuppressive or immunomodulatory therapies.

   - e.g., type 1 juvenile-onset diabetes mellitus, antibody positive for rheumatoid arthritis, Graves disease, Hashimoto thyroiditis, lupus, scleroderma, systemic vasculitis, hemolytic anemia, immune mediated thrombocytopenia, Crohn disease, ulcerative colitis, and psoriasis.
7. Subjects with any known uncontrolled comorbid illness, including ongoing or active infections, symptomatic congestive heart failure (NYHA>2), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Subjects who have received any of the following medications within 4 weeks prior to randomization:

   * Immunotherapy, including monoclonal antibodies, cytokines, interferons, and checkpoint inhibitors.
   * Immunosuppressants, including cyclosporin, rapamycin, tacrolimus, rituximab, alemtuzumab, natalizumab, and cyclophosphamide.
   * Other biologics, including G-CSF and other hematopoietic growth factors.
   * Live attenuated vaccines.
   * IV/oral steroids except single prophylactic use in CT/MRI scan or other one-time use in approved indications. Use of inhaled and topical (except on the injection site) steroids is allowed.
   * Alternative and complementary medicine that may affect the immune system.
   * Other investigational drugs
9. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to Grade 0 or 1 (using National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] version 5.0), except for alopecia and laboratory values listed in the inclusion criteria.
10. Subjects with any known severe allergies (e.g., anaphylaxis) to any active or inactive ingredients in the study drugs.
11. Any other reason that the investigator deems the patient as unsuitable for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival rate | one year
  To evaluate the effect of OBI-833/OBI-821 treatment on improving recurrence-free survival in patients with locally advanced, Globo H-positive esophageal cancer in the adjuvant setting

CONTACTS AND LOCATIONS:
Overall Officials: Jang-Ming Lee, Principal Investigator — Department of Surgery, National Taiwan University Hospital. Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan